CLINICAL TRIAL: NCT03285971
Title: Real-Time Decision Support for Improving Intraoperative Cerebral Perfusion Pressure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Phillip Vlisides, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM117828
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Hypoperfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CPP Alert Group (Experimental): Device: Electronic CPP pager alert anesthesia providers will receive a pager alert when CPP decreases below 60 mmHg (median value over 5-minute epochs)
  Interventions: Other: Electronic CPP pager alert
- Control (No Intervention): This arm will not receive the automated pager alerts.

INTERVENTIONS:
Other: Electronic CPP pager alert — Anesthesia providers will receive a pager alert when CPP decreases beow 60 mmHG (median value over 5-minute epochs)
  Other Names: Alerting system
  Arms: CPP Alert Group

SUMMARY:
Across broad surgical populations, cerebral hypoperfusion is associated with increased mortality, stroke, brain cellular injury, and poor functional outcomes. Based on available evidence, The Brain Trauma Foundation recommends that cerebral perfusion pressure (CPP) be maintained greater than 60 mmHg in high-risk settings to minimize risk of cerebral ischemia. Though several lines of investigation have focused on optimal cerebrovascular management in the intensive care unit and cardiac surgery settings, much less focus has been placed on cerebrovascular management during non-cardiac surgery.

Preliminary data indicate that intraoperative CPP routinely falls below 60 mmHg in neurosurgical and trauma surgery settings, though the relationship between reduced intraoperative CPP and outcomes remains unclear. Furthermore, effective methods by which low intraoperative CPP could be prevented have not been thoroughly investigated, which represents the first required step prior to studying the relationship between intraoperative CPP and clinical outcomes. Thus, the aim of this study is to evaluate the efficacy of an automated algorithm that alerts clinicians to a decrease in CPP below 60 mmHg. This study tests the hypothesis that an automated pager alert system (triggered by CPP falling below 60 mmHg) will increase intraoperative CPP compared to standard of care.

DETAILED DESCRIPTION:
This will be a single-center study taking place at the University of Michigan Health System, Ann Arbor, MI. The study has been approved by the University of Michigan Medical School Institutional Review Board (IRBMED).

Automated pager alert protocols have been previously published from the investigators' department, and this alerting system is used for operational purposes on a daily basis. Surgical patients will be automatically screened using a designed script from the anesthesia information management system (Centricity, Wishahaka, WI).

The script will screen for active surgical patients with intracranial pressure (ICP) data recording in our hospital's non-cardiac operating rooms. When these data are captured, an automated enrollment process will occur if the following electronic charting criteria are met:

* Age ≥ 18 years old
* Case identified as a general anesthetic
* Non-intracranial aneurysm surgery
* Non-pregnant patient

After "anesthetic induction end" time is documented within the case, the alerting system will turn on after a 10-minute grace period. The alerting system will then retroactively measure median CPP values over 5-minute epochs, and if median CPP is < 60 mmHg, the following alphanumeric pager alert will be delivered:

"Patient: LAST NAME, FIRST NAME, OR(N), has a cerebral perfusion pressure < 60 mmHg. Disregard alert for intracranial aneurysm cases or if patient is pregnant."

This alert will be delivered twice total (if criteria are met). The aim of the pager alerts will be to relay information regarding cerebral ischemia risk between when CPP decreases below 60 mmHg. Final clinical decision-making, however, will be left to the anesthesia team. The pager alerts will not otherwise compel action, and no other recommendations will be made.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) surgical patients
* Intracranial pathology requiring intracranial pressure (ICP) monitoring

Exclusion Criteria:

* Intracranial aneurysm surgery
* Cases with pressures monitored from a lumbar drain
* Cardiac surgery cases
* Enrolled in conflicting study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Mean Cerebral Perfusion Pressure (CPP, mmHg) | Assessed intraoperatively for the duration of the CPP monitoring period

SECONDARY OUTCOMES:
Mortality (incidence, %) | Within 30 days of surgery
Postoperative Stroke (incidence, %) | Within 30 days of surgery
Myocardial Infarction (incidence, %) | Within 30 days of surgery
Congestive Heart Failure (incidence, %) | Within 30 days of surgery
Cardiac Dysrythmias (incidence, %) | Within 30 days of surgery
  New onset of any of the following: supraventricular tachycardia, atrial fibrillation, atrial flutter, ventricular fibrilation, ventricular tachycardia, heart block requiring pacing
Acute Respiratory Distress Syndrome, ARDS (incidence, %) | Within 30 days of surgery
Acute Kidney Injury, AKI (incidence, %) | Within 30 days of surgery

OTHER OUTCOMES:
Area Under the Curve (AUC) 60 mmHg (min*mmHg) | Assessed intraoperatively for the duration of the CPP monitoring period
Time Spent with CPP <60 mmHg | Assessed intraoperatively for the duration of the CPP monitoring period
Volume of Cerebrospinal Fluid (CSF) Drained Intraoperatively (mL) | Assessed intraoperatively for the duration of the CPP monitoring period

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Medicine - University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. IX. Cerebral perfusion thresholds. J Neurotrauma. 2007;24 Suppl 1:S59-64. doi: 10.1089/neu.2007.9987. No abstract available. PMID 17511547
- [Background] Moore LE, Sharifpour M, Shanks A, Kheterpal S, Tremper KK, Mashour GA. Cerebral perfusion pressure below 60 mm Hg is common in the intraoperative setting. J Neurosurg Anesthesiol. 2012 Jan;24(1):58-62. doi: 10.1097/ANA.0b013e31822b4f05. PMID 21862931
- [Background] Mashour GA, Tremper KK, Avidan MS. Protocol for the "Michigan Awareness Control Study": A prospective, randomized, controlled trial comparing electronic alerts based on bispectral index monitoring or minimum alveolar concentration for the prevention of intraoperative awareness. BMC Anesthesiol. 2009 Nov 5;9:7. doi: 10.1186/1471-2253-9-7. PMID 19891771
- [Background] Mashour GA, Shanks A, Tremper KK, Kheterpal S, Turner CR, Ramachandran SK, Picton P, Schueller C, Morris M, Vandervest JC, Lin N, Avidan MS. Prevention of intraoperative awareness with explicit recall in an unselected surgical population: a randomized comparative effectiveness trial. Anesthesiology. 2012 Oct;117(4):717-25. doi: 10.1097/ALN.0b013e31826904a6. PMID 22990178
- [Background] Blum JM, Stentz MJ, Maile MD, Jewell E, Raghavendran K, Engoren M, Ehrenfeld JM. Automated alerting and recommendations for the management of patients with preexisting hypoxia and potential acute lung injury: a pilot study. Anesthesiology. 2013 Aug;119(2):295-302. doi: 10.1097/ALN.0b013e3182987af4. PMID 23681144